CLINICAL TRIAL: NCT02179307
Title: Determinants of Intra-individual Variation in Adaptability to Resistance Training of Different Volumes
Brief Title: Individual Response to Different Volumes of Resistance Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inland Norway University of Applied Sciences (Other)
Collaborators: Sykehuset Innlandet HF (Other); Revmatismesykehuset AS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Trainsome 2014#002
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: muscle hypertrophy; strength; resistance training; exercise; physical fitness; health; physical conditioning
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Arm label 1-Set, 3-Set (Experimental): 12-week progressive strength training protocol of different volumes
  Interventions: Behavioral: 12-week progressive strength training protocol

INTERVENTIONS:
Behavioral: 12-week progressive strength training protocol — Every study participant will complete 12 weeks of progressive strength training with one leg performing 1-set per exercise per session and the contralateral leg performing 3-sets per exercise per session. Allocation of dominant/non-dominant leg to either 1- or 3-set protocol will be done in a stratified, randomized fashion (stratified with regard to sex and baseline strength).

SUMMARY:
The literature is not clear as to which training volume to employ during initial phases of resistance training programs to ensure optimal muscular adaptations. The purpose of this study is therefore to compare effects of strength training with low versus moderate volume on muscular function and hypertrophy in previously untrained, healthy individuals. Furthermore, the investigators will relate individual variation in responses to proxy markers of individual training state, such as baseline muscular function and muscle fiber type.

The study will include 25 women and 25 men and will consist of a 12-week resistance training protocol. Each study participant will act as their own control, performing both the low- (1-set) and the moderate-volume (3-sets) protocol, allocated to either the dominant or non-dominant leg, in a stratified and randomized fashion.

Primary outcome measures are thigh muscle cross section area and unilateral knee extension strength. Additionally, muscle fiber type composition will be evaluated as well as additional parameters of muscular function.

The primary hypothesis is that low-volume protocols will be beneficial for individuals with glycolytic muscle phenotypes, whereas the opposite will be true for individuals with more aerobic phenotypes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Non-smoking
* Able to tolerate resistance exercise training

Exclusion Criteria:

* Presence or history of cardiovascular, metabolic, endocrine or neuromuscular disease
* Diagnosed mental health disorder
* Intolerance to local anesthetic
* No experience with exercise training
* Performing regular resistance training (more than 1 session per week during last 12 months)
* Impaired strength/ neuromuscular function due to previous injury
* Recurrent pain in lower back, knee or shoulders
* Taking prescribed medication that may affect outcome of training intervention

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Thigh muscle cross-sectional area | Week 0 (baseline) and 12 (post training intervention)
  Changes in muscle cross sectional area of each thigh from baseline to post intervention, assessed by MRI.
Unilateral knee-extension isometric strength | Week 0 (baseline), 2, 5, 9 (during intervention) and 12 (after training intervention)
  Time course changes in maximum knee extensor, isometric strength evaluated at 120° knee angle (180° fully extended).

SECONDARY OUTCOMES:
Muscle strength | Week 0 (baseline), 2, 5, 9 (during intervention) and 12 (after training intervention)
  Time course changes in maximum isoinertial strength defined by one-repetition maximum in leg press, knee extension, knee flexion, and bench press.
Knee extensors and flexors force-velocity relationship | Week 0 (baseline), 2, 5, 9 (during intervention) and 12 (after training intervention)
  Time course changes in torque measured during maximal voluntary isokinetic contraction at 60°, 120° and 240° ∙ sec-1.
Blood hormonal profiles | Week 0 (baseline), 2 and 12 (post training intervention)
  Resting (week 0, 2 and 12) and acutely exercise-induced (week 2) hormonal profiles (testosterone, insulin-like growth factor 1, growth hormone and cortisol) determined in serum from venous blood samples.
Muscle fiber cross-sectional area | Week 0 (baseline), 2 and 12 (post training intervention)
  Changes in muscle fiber cross-sectional area assessed by immunohistochemistry from muscle biopsy. Determined from muscle biopsy samples (Vastus lateralis).
Protein expression | Week 0 (baseline), 2 and 12 (post training intervention)
  Changes in relative abundance of contractile protein isoforms (myosin heavy chain). Modification of proteins related to muscle hypertrophy in relation to an acute exercise session (assessed during week 2 of the intervention). Determined from muscle biopsy samples (Vastus lateralis).
Gene expression | Week 0 (baseline), 2 and 12 (post training intervention)
  Changes in gene expression related to skeletal muscle hypertrophy and structural phenotype measured in steady state conditions (biopsy sampled in resting conditions, week 0, 2 and 12) and in relation to acute exercise (biopsy sampled 1-h after strength exercise, week 2). Determined from muscle biopsy samples (Vastus lateralis).

OTHER OUTCOMES:
Body composition changes | Week 0 (baseline) and 12 (post training intervention)
  Changes in body compositions (lean mass and fat mass) from prior intervention to after intervention assessed by dual x-ray absorptiometry scan.
Habitual physical activity | Week 0
  Self-reported prior habitual physical activity assessed by questionnaire and interview before training intervention
Daily nutrient intake | Week 6
  Daily nutrient intake assessed by a 4-day food intake registration.

CONTACTS AND LOCATIONS:
Overall Officials: Stian Ellefsen, PhD, Principal Investigator — Inland Norway University of Applied Sciences
Locations (1):
- Lillehammer University College, Lillehammer, Norway